CLINICAL TRIAL: NCT00464919
Title: A Phase II Study of Sorafenib Plus Tegafur/Uracil for the Treatment of Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: Sorafenib Plus Tegafur/Uracil (UFUR®) for Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chih-Hung Hsu, Department of Oncology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 950914
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Advance, hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Tegafur; Uracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: Sorafenib; Drug: tegafur/uracil (UFUR®)

INTERVENTIONS:
Drug: Sorafenib
Drug: tegafur/uracil (UFUR®)

SUMMARY:
The prognosis for patients with metastatic or locally advanced hepatocellular carcinoma (HCC) is poor. The role of conventional systemic chemotherapy has been very limited because most chemotherapeutic agents are in-effective and relative toxic to HCC patients who tend to have poor organ function reserves due to liver cirrhosis. The molecular-targeted therapy, which aims at deranged signaling pathways of cancer cells or their microenvironment, holds promise for HCC.

Sorafenib (BAY 43-9006), a novel bi-aryl urea, is a potent inhibitor of VEGFR2 and Raf kinase. The clinical activity of sorafenib in HCC has been tested in a phase II study (Bayer study 10874), which enrolled a total of 137 advanced HCC patients. There were 4% of documented partial response, 5% of minor response, and 55% of stable disease. The 6- month progression -free for the cohort was 40%. Currently, there are two on-going large-scale randomized trials of sorafenib in advanced HCC patients worldwide.

DETAILED DESCRIPTION:
The prognosis for patients with metastatic or locally advanced hepatocellular carcinoma (HCC) is poor. The role of conventional systemic chemotherapy has been very limited because most chemotherapeutic agents are in-effective and relative toxic to HCC patients who tend to have poor organ function reserves due to liver cirrhosis. The molecular-targeted therapy, which aims at deranged signaling pathways of cancer cells or their microenvironment, holds promise for HCC.

Sorafenib (BAY 43-9006), a novel bi-aryl urea, is a potent inhibitor of VEGFR2 and Raf kinase. The clinical activity of sorafenib in HCC has been tested in a phase II study (Bayer study 10874), which enrolled a total of 137 advanced HCC patients. There were 4% of documented partial response, 5% of minor response, and 55% of stable disease. The 6- month progression -free for the cohort was 40%. Currently, there are two on-going large-scale randomized trials of sorafenib in advanced HCC patients worldwide.In this study proposal, we propose to combine sorafenib with metronomic chemotherapy in the treatment of advanced HCC patients. It has been recently demonstrated that cytotoxic chemotherapy, when given in a low-dose, continuous, and uninterrupted way (i.e. the "metronomic" chemotherapy), inhibits tumor angiogenesis. The anti-angiogenesis effect of metronomic chemotherapy can be potentiated by combining the inhibitors of VEGF/VEGFR pathway. UFUR®, a composite drug composed of tegafur and uracil, is an orally active 5-fluorouracil (5-FU) preparation. The activity of tegafur/uracil in HCC has been tested in two relatively small-scale phase II studies, with objective tumor response rates ranging from 0~18%. Interestingly, tegafur and its metabolites, including γ-hydroxybutyric acid and γ-butyrolactone, have been shown to be potent inhibitors of angiogenesis in several preclinical models. Therefore, tegafur/uracil (UFUR®), which has potential anti-HCC activity and interesting anti-angiogenesis activity, is an ideal candidate drug to improve the efficacy of sorafenib in HCC.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* ECOG PS 0-2;
* Histologically or cytologically documented unresectable and/or metastatic HCC;
* Measurable disease by RECIST criteria;
* Previous local therapy completed > 6 weeks;
* Any acute toxicity (CTC-AE) < grade 1;
* Child-Pugh A;
* Liver transaminases ≤ 5 x ULN;
* Albumin ≥ 2.8 g/dl;
* Serum total bilirubin ≤ 3 mg/dl;
* INR ≤ 2.3 or PT ≤ 6 seconds above control;
* WBC ≥ 3,000/µl;
* ANC ≥ 1,500/µl;
* Platelets ≥ 100,000/µl;
* Hb ≥ 8.5 g/dl;
* Creatinine ≤ 1.5 x ULN; AND
* Amylase and lipase < 1.5 x ULN

Exclusion Criteria:

* Metastatic brain/leptomeningeal tumors;
* Prior or concomitant systemic anti-cancer treatment for HCC, including:

  * Systemic chemotherapy (TACE is allowed)
  * Immunotherapy
  * Hormonal therapy (hormonal therapy used for supportive used is allowed)
  * Raf-kinase inhibitors
  * MEK inhibitors
  * Farnesyl transferase inhibitors
  * VEGF/VEGFR- inhibitors or other anti-angiogenesis agents
  * Investigational anti-cancer agents
* Severe and/or uncontrolled medical conditions:

  * Uncontrolled high blood pressure
  * History of poor compliance with anti-hypertensive agents
  * Active or uncontrolled infection
  * Unstable angina
  * CHF
  * MI or CVA < 6 months
  * GI bleeding < 30 days
  * Unable to take oral medications
* Severe renal impairment which requires dialysis; proteinuria > grade 2;
* BMT or stem cell rescue < 4 months; organ transplant;
* HIV infection;
* Major surgical procedure, open biopsy, or significant traumatic injury < 4 weeks or those who receive minor surgical procedures (e.g. core biopsy or fine needle aspiration) within 2 weeks;
* Receive central venous line placement within 7 days;
* Patients who anticipate receiving major surgery during the course of the study;
* Use rifampin, St. John's Wort [Hypericum perforatum];
* Patients taking narrow therapeutic index medications will be monitored closely. These include warfarin, phenytoin, quinidine, carbamazepine, phenobarbital, cyclosporine, and digoxin; OR
* Patients for whom tegafur is contra-indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-04; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine the progression- free survival of sorafenib plus tegafur/uracil (UFUR®) for the treatment of advanced or metastatic HCC. | 2007~2008

SECONDARY OUTCOMES:
The 6-month progression-free survival rate. | 2007~2008
The objective tumor response rate. | 2007~2008
The disease stabilization rate (complete response + partial response + stable disease for at least 2 months). | 2007~2008
The overall survival. | 2007~2008
The safety profile. | 2007~2008
To evaluate the changes of circulating biomarkers indicating the angiogenesis activity and their correlation with objective tumor response. | 2007~2008

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Hsu, M.D.Ph.D, Study Chair — Department of Oncology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hsu CY, Shen YC, Yu CW, Hsu C, Hu FC, Hsu CH, Chen BB, Wei SY, Cheng AL, Shih TT. Dynamic contrast-enhanced magnetic resonance imaging biomarkers predict survival and response in hepatocellular carcinoma patients treated with sorafenib and metronomic tegafur/uracil. J Hepatol. 2011 Oct;55(4):858-65. doi: 10.1016/j.jhep.2011.01.032. Epub 2011 Feb 19. PMID 21338641